CLINICAL TRIAL: NCT03333304
Title: A Randomized Prospective Clinical Trial to Assess the Role of Procalcitonin-guided Antimicrobial Therapy to Reduce Long-term Infections Sequelae
Brief Title: A Clinical Trial of Procalcitonin-guided Antimicrobial Therapy in Sepsis
Acronym: PROGRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROGRESS
Record Dates: First submitted 2017-10-23; First posted 2017-11-06 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Sepsis
Keywords: Procalcitonin
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized at 1:1 ratio by a separate list per study site into two treatment groups. The two groups of treatment will be as follows:
  * Standard of care: these patients will receive antimicrobials according to standard practice of the attending physicians but PCT will not be measured and antimicrobials will be stopped according to the local standard practice.
  * PCT group: these patients will receive antimicrobials according to standard practice of the attending physicians and antimicrobials will be discontinued according to PCT kinetics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCT group (Experimental): Procalcitonin measurement and Discontinuation of antimicrobials according to Procalcitonin kinetics
  Interventions: Diagnostic Test: Procalcitonin measurement
- Standard of care (No Intervention): Standard practice

INTERVENTIONS:
Diagnostic Test: Procalcitonin measurement — Discontinuation of antimicrobials according to Procalcitonin Kinetics
  Arms: PCT group

SUMMARY:
The aim of the study is to demonstrate if using one procalcitonin (PCT)-guided rule of stop of antimicrobials, the incidence of infections by C.difficile and by Multi-Drug-Resistant (MDR) bacteria during the next six months may be significantly decreased.

DETAILED DESCRIPTION:
Early administration of antimicrobials remains the mainstay of treatment of severe infections. Current guidelines of management of severe sepsis suggest that initial therapy of a patient should be reviewed after 48 to 72 hours. At that stage some patients are doing well, whereas others fail to respond. When microbiology cultures of biological specimens fail to provide information for the microbial cause of an infection and susceptibilities to antimicrobials, antimicrobial stewardship relies on the use of biomarkers and mainly procalcitonin (PCT). Data so far, suggest that early changes of serum PCT can inform about the prognosis of the septic patient, with greater values reflecting a worse outcome and higher mortality and that serial measurements within 48-72 hours provide adequate information of the appropriateness of the administered antimicrobials. Moreover the use of a procalcitonin guided-treatment in surgical as well as in non-surgical critically-ill patients, is seen to be non-inferior to the standard antibiotic approach and leads to a shorter antibiotic exposure, having possible beneficial effect on reducing microbial resistance and therapy costs.

In the largest study conducted so far, de Jong et al showed that PCT-guided stop of treatment was not only safe compared with standard of care antibiotic duration, but also led to a better outcome i.e. significant decrease of both 28-day and 1-year mortality. The results of this study are a major contribution in the field of critical care since they prove for the first time that PCT guidance of antimicrobial treatment allows not only proper antimicrobial stewardship but it is also associated with survival benefit. However, de Jong et al did not provide findings to explain the underlying mechanism of survival benefit. As a rule critically ill patients run two major risks coming from the long-term administration of antimicrobials; the first is infections by Clostridium difficile coming from the ecological damage of gut flora and the second is the risk of infections by multidrug-resistant (MDR) bacteria colonizing the gut. MDR is emerging after the ecological pressure of broad-spectrum antimicrobial usually administered to the critically ill patient.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* In case of women, unwillingness to remain pregnant during the study period.
* Age more than or equal to 18 years
* Sequential Organ Failure Assessment (SOFA) score more than or equal to 2 points for patients admitted in the emergencies and with a more than or equal to a 2-point increase of admission SOFA score for hospitalized patients.
* Presence of one of the following infections: community-acquired pneumonia, hospital-acquired pneumonia, ventilator-associated pneumonia, bacteremia and acute pyelonephritis. Any infection with onset more than 48 hours post hospital admission is considered one hospital-acquired infection.

Exclusion Criteria:

* Failure to obtain written consent to participate
* Patients in pregnancy or breastfeeding. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study
* Patients receiving prolonged antibiotic therapies ( e.g. endocarditis, implantable device-associated infection, cerebral/hepatic abscess, osteomyelitis, meningitis)
* Patients with severe infections due to viruses or parasites (e.g. Dengue, Toxoplasma gondii, Plasmodium spp.)
* Patients infected with Mycobacterium tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
The change of infection-associated adverse events rate. The infection-associated adverse events rate are any case of Clostridium Difficile Infection (CDI) or infection by MDR or infection-related death. | 6 months
  The change of infection-associated adverse events rate. The infection-associated adverse events rate are any case of Clostridium Difficile Infection (CDI) or infection by MDR or infection-related death.

SECONDARY OUTCOMES:
Infection-associated adverse events rate | 6 months
  Time to first infection-associated adverse events rate
Clostridium difficile Infection | 6 months
  Rate of infections by Clostridium difficile
Infections by MDR | 6 months
  Rate of infections by MDR
Mortality | 28 days
  Mortality
Mortality | 6 months
  Mortality
Stool colonization by C.difficile | 6 months
  Rate stool positive for GDH by C.difficile
Stool colonization by MDR | 6 months
  Rate of stool colonization by MDR
Microbiome composition | 28 days
  Microbiome composition
Changes of the microbiome | 28 days
  Changes of the microbiome
Consumption of antimicrobials during hospitalization | 28 days
  Consumption of antimicrobials during hospitalization
Cost of hospitalization | 28 days
  Real cost of hospitalization i.e medicines administered and interventions performed, in Euro, between the two groups of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Antoniadou, MD, PhD, Principal Investigator — National Kapodistrian University of Athens, Medical School
Locations (7):
- Greece (7):
  - 1st Department of Internal Medicine, General Hospital of Athens "G. Gennimatas", Athens
  - 3rd Department of Internal Medicine, Sotiria Athens General Hospital, Athens
  - 4th Department of Internal Medicine, Attikon University Hospital, Athens
  - 2nd Department of internal Medicine, General Hospital of Attiki "Sismanogleio", Athens
  - 1st Department of Internal Medicine, General Hospital of Elefsina "Thriasio", Athens
  - 2nd Department of Internal Medicine, General Hospital of Elefsina "Thriasio", Athens
  - 2nd Department of Internal Medicine, General Hospital of Piraeus "Tzaneio", Piraeus

REFERENCES:
- [Derived] Kyriazopoulou E, Stylianakis E, Damoraki G, Koufargyris P, Kollias I, Katrini K, Drakou E, Marousis K, Spyrou A, Symbardi S, Alexiou N, Alexiou Z, Lada M, Poulakou G, Chrysos G, Adamis G, Giamarellos-Bourboulis EJ. Procalcitonin-guided early cessation of antibiotics prevents gut inflammation and preserves gut microbiome: Data from the PROGRESS controlled trial. Int J Antimicrob Agents. 2025 Aug;66(2):107507. doi: 10.1016/j.ijantimicag.2025.107507. Epub 2025 Apr 9. PMID 40216091
- [Derived] Kyriazopoulou E, Karageorgos A, Liaskou-Antoniou L, Koufargyris P, Safarika A, Damoraki G, Lekakis V, Saridaki M, Adamis G, Giamarellos-Bourboulis EJ. BioFire(R) FilmArray(R) Pneumonia Panel for Severe Lower Respiratory Tract Infections: Subgroup Analysis of a Randomized Clinical Trial. Infect Dis Ther. 2021 Sep;10(3):1437-1449. doi: 10.1007/s40121-021-00459-x. Epub 2021 Jun 13. PMID 34120316
- [Derived] Kyriazopoulou E, Liaskou-Antoniou L, Adamis G, Panagaki A, Melachroinopoulos N, Drakou E, Marousis K, Chrysos G, Spyrou A, Alexiou N, Symbardi S, Alexiou Z, Lagou S, Kolonia V, Gkavogianni T, Kyprianou M, Anagnostopoulos I, Poulakou G, Lada M, Makina A, Roulia E, Koupetori M, Apostolopoulos V, Petrou D, Nitsotolis T, Antoniadou A, Giamarellos-Bourboulis EJ. Procalcitonin to Reduce Long-Term Infection-associated Adverse Events in Sepsis. A Randomized Trial. Am J Respir Crit Care Med. 2021 Jan 15;203(2):202-210. doi: 10.1164/rccm.202004-1201OC. PMID 32757963